CLINICAL TRIAL: NCT05920265
Title: Quadratus Lumborum Plain Block Versus Fascia Iliac Block in Hip Fracture
Brief Title: Quadratus Lumborum Plain Block Versus Fascia Iliac Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hassan Mokhtar Elshorbagy Hetta, lecturer of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16:2021
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Post Operative Pain
Keywords: QLB; Fascia Iliac Block; hip surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quadratus Lumborum Block (Experimental)
  Interventions: Procedure: Quadratus Lumborum plain Block
- Fascia Iliac Block (Experimental)
  Interventions: Procedure: fascia iliaca block
- control (Active Comparator)
  Interventions: Diagnostic Test: control group

INTERVENTIONS:
Procedure: Quadratus Lumborum plain Block — ultrasound guided Quadratus Lumborum plain Block using 0.5 ml/kg bupivacaine 0.25% .
  Arms: Quadratus Lumborum Block
Procedure: fascia iliaca block — ultrasound guided fascia iliaca block using 0.5 ml/kg bupivacaine 0.25%
  Arms: Fascia Iliac Block
Diagnostic Test: control group — no intervention
  Arms: control

SUMMARY:
evaluation the efficacy of Quadratus Lumborum plain Block Versus Fascia Iliac Block for postoperative pain after hip surgery

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years
* fracture hip

Exclusion Criteria:

* patients refuse
* mental problem patient with any coagulation deficiency or bleeding problems patient with allergy to investigated medications,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
analgesic consumption | 24 hour
  intraoperative and post operative

SECONDARY OUTCOMES:
Visual analogue pain score | 24 hour
  score 0-10 which mean 0 no pain and 10 the worst pain
first analgesic demand | 24 hour
  the first time to intake rescue analgesia

CONTACTS AND LOCATIONS:
Overall Officials: abeer M hassaneen, Ass. professor, Study Director — minia university hospital/ faculty of medicine; ahmed H Mohamed, Professor, Study Chair — minia university hospital/ faculty of medicine
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No